CLINICAL TRIAL: NCT05922644
Title: The Safety and Efficacy of Short-term Cervical Spinal Cord Stimulation in Patients With Disorders of Consciousness After Intracerebral Hemorrhage: a Multicenter, Prospective, Randomized, Outcome-blind Interventional Study
Brief Title: Short-term Cervical Spinal Cord Stimulation in Patients With Disorders of Consciousness After Intracerebral Hemorrhage
Acronym: SCS-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Rehabilitation Hospital Affiliated to National Research Center for Rehabilitation Technical Aids (Unknown); Shenzhen Qianhai Shekou Free Trade Zone Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Yong Cao, director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022GKZS0005
Record Dates: First submitted 2023-05-25; First posted 2023-06-28 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Coma; Stroke
MeSH Terms: conditions — Coma; Stroke | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal cord electrical stimulation group (Experimental): According to the EDC system, patients are randomly assigned to receive 21 days of cervical spinal cord electrical stimulation treatment in addition to routine brain resuscitation and rehabilitation awakening treatment.
  Interventions: Device: SCS
- Conventional treatment group (Sham Comparator): According to the EDC system, patients are randomly assigned to receive only routine brain resuscitation and rehabilitation awakening treatment.
  Interventions: Other: Conventional

INTERVENTIONS:
Device: SCS — 21 days of cervical spinal cord electrical stimulation treatment in addition to routine brain resuscitation and rehabilitation awakening treatment.
  Arms: Spinal cord electrical stimulation group
Other: Conventional — Routine brain resuscitation and rehabilitation awakening treatment.
  Arms: Conventional treatment group

SUMMARY:
Disorders of consciousness (DOC) refers to the persistent loss of consciousness after 28 days in patients with brain injury caused by trauma, stroke, or hypoxia. It includes coma, vegetative state, and minimally conscious state. At present, there is no effective treatment for DOC. Only one RCT study of amantadine has proved that it may be effective for the treatment of DOC. In recent years, more evidence has shown that neuromodulation technology is beneficial to the recovery of DOC. Cervical spinal cord stimulation surgery is a new treatment method for patients with DOC. Electrodes are implanted in the high cervical spinal cord C2-C5. By adjusting different electrical stimulation parameters, it has a wake-promoting effect. In this study, patients were selected into the spinal cord stimulation group and the conventional treatment group according to the wishes of their families. The patients in the spinal cord stimulation group were given 21 days of cervical spinal cord stimulation treatment on the basis of conventional brain rehabilitation. Patients were followed up routinely and completed designated examinations at 12 months to determine the safety and efficacy of cervical spinal cord stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Patients with postoperative consciousness disorders after cerebral hemorrhage for more than 28 days
* CRS-R score meets the MCS diagnosis
* Signed informed consent.

Exclusion Criteria:

* Secondary brain injury caused by arteriovenous malformation, cerebral aneurysm, cavernous hemangioma, brain tumor and carbon monoxide poisoning
* History of previous epileptic seizures
* Critical condition, unstable intracranial condition, risk of rebleeding
* Unstable vital signs requiring mechanical ventilation
* Contraindications for spinal cord surgery
* Severe sympathetic overactivity syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in consciousness 12 months after surgery assessed by CRS-R | 12 months
  The primary efficacy indicator is "change in consciousness recovery 12 months after cervical spinal cord electrical stimulation (assessed by the Coma Recovery Scale - Revised (CRS-R), ranges from 0 to 25, with higher scores mean a better outcome)".

SECONDARY OUTCOMES:
Consciousness recovery 12 months after surgery assessed by GOS-E | 12 months
  The secondary efficacy indicator is "consciousness recovery 12 months after surgery (assessed by the Glasgow Outcome Scale - Extended (GOS-E) to evaluate the patient's consciousness status, ranges from 0 to 8, with higher scores mean a better outcome)".

OTHER OUTCOMES:
Glasgow Coma Scale (GCS) | 12 months
  Exploratory Indicators, ranges from 0 to 15, with higher scores mean a better outcome.
National Institute of Health stroke scale (NIHSS) | 12 months
  Exploratory Indicators, ranges from 0 to 42, with higher scores mean a worse outcome.
Full Outline of UnResponsiveness (FOUR) Score | 12 months
  Exploratory Indicators, ranges from 0 to 16, with higher scores mean a better outcome.
Disability rating scale (DRS) | 12 months
  Exploratory Indicators, ranges from 0 to 29, with higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided